CLINICAL TRIAL: NCT05892939
Title: Effects of Intranasal Oxytocin on Fear Processing in Naturalistic Contexts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-BAM-06
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Oxytoxin; Fear; Social; fMRI

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytoxin group (Experimental): Drug: intranasal Oxytocin(24IU)
  Interventions: Drug: intranasal Oxytocin(24IU)
- Placebo group (Placebo Comparator): Drug: intranasal Placebo
  Interventions: Drug: intranasal Placebo

INTERVENTIONS:
Drug: intranasal Oxytocin(24IU) — Administration of intranasal Oxytocin(24IU)
  Arms: Oxytoxin group
Drug: intranasal Placebo — Administration of intranasal Placebo
  Arms: Placebo group

SUMMARY:
The main aim of the study is to investigate the modulatory effects of intranasal oxytocin (24IU) on fear in naturalistic social and non-social contexts and the underlying neural mechanisms.

DETAILED DESCRIPTION:
In a double-blind placebo-controlled between-subject experimental design, 60 adult male subjects will be randomly allocated to receive either intranasal oxytocin (24IU, n= 30) or placebo (n = 30) nasal spray. 45 minutes after treatment the participants will undergo a naturalistic fear induction paradigm during fMRI. During the paradigm video clips of 25s lengths will be presented showing fear-inducing situations in social and non-social contexts as well as corresponding control video clips. Following each clip subjects are required to rate their level of subjective fear on a rating scale ranging from 1 (no fear) to 9 (highest fear). Participants will undergo screening for psychopathological and emotional states before treatment. Together with a randomized assignment to the treatment groups, this will allow controlling for confounding between-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness
* Normal or corrected-normal version

Exclusion Criteria:

* History of head injury
* Medical or psychiatric illness
* Hypertension
* General cardio-vascular alteration or diseases
* Allergy against medications
* Visual or motor impairments
* Claustrophobia
* Drug addiction
* Nicotine dependence
* FMRI contradictions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
BOLD-level activity as assessed by functional magnetic resonance imaging (fMRI) | 45 minutes to 70 minutes after treatment
  BOLD-level activity as assessed by functional magnetic resonance imaging (fMRI) in response to four conditions of movie clips (Fear-Social\FS, Fear-Non-social\FNS, Neutral-Social\NS, Neutral-Non-social\NNS). Effects of Oxytocin on the neural basis of fear will be examined by comparing the treatment groups (Oxytocin versus Placebo) with respect to fearful versus non fearful conditions. The investigators expect that Oxytocin will decrease reactivity in emotion reactive brain regions as compared to Placebo.

SECONDARY OUTCOMES:
Experienced fear during the paradigm as assessed by self-reported ratings | 45 minutes to 70 minutes after treatment
  Experienced fear during the paradigm as assessed by self-reported ratings on a 1-9 point Likert-scale ranging from 1 (no fear) to 9 (highest fear). Participants will rate their subjective level of fear following each video clip. Effects of Oxytocin on the level of subjective fear will be examined by comparing the treatment groups (Oxytocin versus Placebo) with respect to the self-reported fear levels. The investigators expect that Oxytocin will decrease the level of subjective fear experience compared to Placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China